CLINICAL TRIAL: NCT06275243
Title: Alzheimer's Disease as a Sociosanitary Priority: ApoE Gene Polymorphism
Brief Title: Polymorphism of ApoE in Alzheimer's Disease: Genetic Study in Castile and Leon (Spain)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de León (Other)
Collaborators: Consejo General de Colegios Oficiales de Enfermería España (Unknown)
Responsible Party: Principal Investigator, Leticia Sánchez Valdeón, Assistant Professor Doctor in University of León, Universidad de León
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ETICA-ULE-021-2022
Record Dates: First submitted 2024-01-30; First posted 2024-02-23 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease; ApoE polymorphism; Geographical distribution; Cardiovascular factors; Total cholesterol
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: It is a longitudinal randomised clinical study, in which two study groups were used. A group of cases diagnosed with Alzheimer's disease and a control group of healthy individuals without Alzheimer's disease.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of cases diagnosed with Alzheimer's disease (Active Comparator): Participants: Men and women with age between 60 and 90 years
  Interventions: Diagnostic Test: Kit Buccal swab collection & stabilization de Canvax®; Other: Cholesterol levels according to ApoE Genotype; Other: Assessing cardiovascular risk factors in all participants
- Control group of healthy individuals without a diagnosis of Alzheimer's disease (Sham Comparator): Participants: Men and women with age between 60 and 90 years
  Interventions: Diagnostic Test: Kit Buccal swab collection & stabilization de Canvax®; Other: Assessing cardiovascular risk factors in all participants

INTERVENTIONS:
Diagnostic Test: Kit Buccal swab collection & stabilization de Canvax® — Assessment of ApoE variant in saliva samples as a potential biomarker for Alzheimer's disease.
Other: Cholesterol levels according to ApoE Genotype — Enhancing the quality of life of study participants by investigating cholesterol levels based on their ApoE genotype.
  Arms: Group of cases diagnosed with Alzheimer's disease
Other: Assessing cardiovascular risk factors in all participants — Through individual interviews, record cardiovascular factors and assess their correlation with Alzheimer's disease.

SUMMARY:
The general objective of this randomized and longitudinal clinical study was to estimate the frequencies of ApoE variants both in the user population of the "Messengers of Peace" Residences and the "Associations of Relatives of Alzheimer's Patients" in Castile y Leon, since, due to its geographical location at the crossroads, it has received multiple genetic contributions from both northern Europe, the Mediterranean area and northern Africa.

The main questions it aims to answer are:

* What are the allelic frequencies of ApoE variants in the population of individuals with Alzheimer's disease in Castile and Leon?
* Is there a correlation between the ApoE4 variant and the lipid profile in the blood of individuals with Alzheimer's disease in this region?

DETAILED DESCRIPTION:
In the context of Alzheimer disease research, it is widely recognized that the ApoE gene plays a fundamental role in the genetic predisposition of this disease. With three major alleles: ApoE2, ApoE3, and ApoE4, genetic variability in the ApoE gene has been the subject of extensive attention in previous research and its association with increased risk of Alzheimer's disease has remained consistent. Within this framework, three hypotheses are proposed focused on understanding the specific influence of ApoE on Alzheimer's disease and exploring the possible underlying mechanisms.

Within this framework, three hypotheses are proposed focused on understanding the specific influence of ApoE on Alzheimer disease and exploring the possible underlying mechanisms:

1. - Research hypotheses: The genetic variant ApoE4/4 is significantly related to a higher risk of developing Alzheimer's disease compared to individuals who do not carry this genotype.
2. - Research hypotheses: The ApoE2/2 genetic variant is associated with a lower risk of developing Alzheimer's disease compared to other genotypes.
3. - Research hypotheses: People who carry the ApoE4 isoform have elevated levels of total cholesterol and LDL-cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Be between 60 and 90 years old.
* Subjects with a diagnosis of AD in the case group.
* Subjects free of AD diagnosis in the control group.
* Subjects who voluntarily and consented to participate free of charge.
* Have completed the written consent

Exclusion Criteria:

* Subjects who, at the time of sample collection, had behavioral or other alterations that made the sample collection procedure impossible.
* Subjects who, at the time of sample collection, presented oral alterations incompatible with the technique.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Distribution of ApoE variants in the Alzheimer's disease population diagnosed in Castile and Leon. | 9 months
  The saliva samples will be processed to purify and extract DNA. Subsequently, a PCR amplification will be performed to check the ApoE alleles and genotypes.

SECONDARY OUTCOMES:
Cardiovascular factors in individuals with Alzheimer's disease and healthy subjects. | 9 months
  We will analyze whether there are significant differences between individuals with Alzheimer's disease and healthy subjects in terms of cardiovascular risk factors (Diabetes mellitus, cardiac pathology, hypercholesterolemia and high blood pressure) using the z-test for difference in proportions.
ApoE genotypes and cholesterol levels in the Alzheimer's disease population diagnosed in Castile and Leon. | 9 months
  To assess the presence of significant differences in the mean cholesterol values across different genotypes, an analysis of variance (ANOVA) test will be applied.

CONTACTS AND LOCATIONS:
Locations (1):
- University of León, León, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alharbi KK, Syed R, Alharbi FK, Khan IA. Association of Apolipoprotein E Polymorphism with Impact on Overweight University Pupils. Genet Test Mol Biomarkers. 2017 Jan;21(1):53-57. doi: 10.1089/gtmb.2016.0190. PMID 28085496
- [Background] Pantelidis P, Lambert-Hammill M, Wierzbicki AS. Simple sequence-specific-primer-PCR method to identify the three main apolipoprotein E haplotypes. Clin Chem. 2003 Nov;49(11):1945-8. doi: 10.1373/clinchem.2003.021683. No abstract available. PMID 14578332
- [Background] Reales G, Hernandez CL, Dugoujon JM, Novelletto A, Cuesta P, Fortes-Lima C, Rodriguez JN, Calderon R. New insights into the distribution of APOE polymorphism in the Iberian Peninsula. The case of Andalusia (Spain). Ann Hum Biol. 2014 Sep-Oct;41(5):443-52. doi: 10.3109/03014460.2013.877966. Epub 2014 Feb 6. PMID 24502694
- [Background] Eisenberg DT, Kuzawa CW, Hayes MG. Worldwide allele frequencies of the human apolipoprotein E gene: climate, local adaptations, and evolutionary history. Am J Phys Anthropol. 2010 Sep;143(1):100-11. doi: 10.1002/ajpa.21298. PMID 20734437
- [Background] Reitz C, Mayeux R. Use of genetic variation as biomarkers for Alzheimer's disease. Ann N Y Acad Sci. 2009 Oct;1180:75-96. doi: 10.1111/j.1749-6632.2009.04945.x. PMID 19906263
- [Background] Salameh TS, Rhea EM, Banks WA, Hanson AJ. Insulin resistance, dyslipidemia, and apolipoprotein E interactions as mechanisms in cognitive impairment and Alzheimer's disease. Exp Biol Med (Maywood). 2016 Sep;241(15):1676-83. doi: 10.1177/1535370216660770. Epub 2016 Jul 28. PMID 27470930
- [Background] Gonzalez RD, Gomes I, Gomes C, Rocha R, Duraes L, Sousa P, Figueruelo M, Rodriguez M, Pita C, Hornero R, Gomez C, Lopes AM, Pinto N, Martins S. APOE Variants in an Iberian Alzheimer Cohort Detected through an Optimized Sanger Sequencing Protocol. Genes (Basel). 2020 Dec 22;12(1):4. doi: 10.3390/genes12010004. PMID 33375167